CLINICAL TRIAL: NCT03371615
Title: A Randomised, Controlled, Double Blind Trial to Evaluate the Tolerance and Safety of a New Partly Fermented Anti-regurgitation Infant Formula Containing Prebiotics and Locust Bean Gum in Infants With Regurgitation.
Brief Title: Evaluation of the Tolerance and Safety of a New Partly Fermented Anti-regurgitation Infant Formula
Acronym: Leopard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBB16GL10424
Record Dates: First submitted 2017-10-24; First posted 2017-12-13 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2019-11

CONDITIONS: Regurgitation, Gastric
MeSH Terms: conditions — Laryngopharyngeal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fermented IF + LBG + Gos Fos (Active Comparator): Fermented infant formula with Locust bean gum and Gos Fos
  Interventions: Other: Anti-regurgitation infant formula
- Fermented IF +LBG (Placebo Comparator): Fermented infant formula with Locust bean gum
  Interventions: Other: Anti-regurgitation infant formula

INTERVENTIONS:
Other: Anti-regurgitation infant formula — Anti regurgitation infant formula

SUMMARY:
A randomised, controlled, double-blind trial to evaluate the tolerance and safety of a new partly fermented anti-regurgitation infant formula containing prebiotics and locust bean gum in infants with regurgitation.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton healthy term infant aged 3 - 13 weeks;
2. Gestational age at birth 37- 42 weeks;
3. Normal birth weight for gestational age and gender i.e. 10th to 90th percentile compared to the WHO or local growth charts;
4. Infants with regurgitation that are otherwise healthy, based upon the following criteria: 1) Regurgitation of 2 or more times per day for 1 or more weeks according to reported history, 2) an indication for the use of AR formula according to the investigator at screening/randomisation.
5. Fully formula fed for at least 7 days before screening/randomisation;
6. Written informed consent from the parent(s) and/or legally acceptable representative(s), aged ≥ 18 years.

   -

Exclusion Criteria:

* 1. History of retching, hematemesis, aspiration, apnoea, failure to thrive, feeding or swallowing difficulties or abnormal posturing; 2. Gastrointestinal infection within 4 weeks prior to randomisation; 3. Congenital condition and/or previous or current illness and (or) medication use that could interfere with the main study outcomes according to the investigator; 4. Known cow's milk protein allergy, lactose intolerance, or galactosaemia including history of any other allergic manifestations or known allergy to any of the study product ingredients (especially scGOS); 5. Presence of any other gastrointestinal symptom(s)/disorder(s) that are not functional in nature, as assessed by the investigator's clinical judgement; 6. Received any of the following products/medication prior to randomisation: systemic antibiotics, prokinetics, proton pump inhibitors, complementary feeding/weaning within 4 weeks prior to randomisation; 7. Incapability of the parent(s) to comply with the study protocol or investigator's uncertainty about the willingness or ability of the parent(s) to comply with the protocol requirements; 8. Current participation in another clinical intervention study.

Ages: 3 Weeks to 13 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2017-11-04 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
GI tolerance | 4 weeks
  To assess the gastrointestinal (GI) tolerance of the investigational product compared to the control product based on Infant Gastrointestinal Symptom Questionnaire(IGSQ) symptoms score containg 13 questions on a 7 point scale

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Poliklinika Ginekologiczno-Poloznicza Sp. Z.O.O Sp.K, Bialystok
  - Centrum Medyczne Promed, Krakow

REFERENCES:
- [Background] Bellaiche M, Ludwig T, Arciszewska M, Bongers A, Gomes C, Swiat A, Dakhlia F, Piollet A, Oozeer R, Vandenplas Y. Safety and Tolerance of a Novel Anti-Regurgitation Formula: A Double-Blind, Randomized, Controlled Trial. J Pediatr Gastroenterol Nutr. 2021 Nov 1;73(5):579-585. doi: 10.1097/MPG.0000000000003289. PMID 34417399